CLINICAL TRIAL: NCT04301167
Title: Loneliness and Health: The Moderating Role of Befriending Services
Acronym: HALO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Queen's University, Belfast (Other); Newcastle University (Other); University of Limerick (Other); St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Joanna McHugh, Adjunct Assistant Professor, University of Dublin, Trinity College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APA2017004
Record Dates: First submitted 2020-02-25; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Loneliness
Keywords: brain health; loneliness; aging; quality of life

STUDY DESIGN:
Intervention Model Description: AB single-case experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): An AB single-case experimental design will be used. An RCT would be inappropriate since the befriending intervention is known to improve wellbeing. As such participants will have data collected in a pre- and post-intervention phase, for a maximum of 13 time points. This approach has been identified by What Works Clearinghouse as an acceptable empirical design to include in evidence based practice reviews (Kratchowill et al., 2010).
  Interventions: Behavioral: befriending

INTERVENTIONS:
Behavioral: befriending — Participants are new users of the ALONE befriending intervention, which matches participants to volunteer befrienders who visit once weekly for a minimum of 12 months. It is a criterion of study involvement that participants commit to completing at least two data collection timepoints before being matched to a befriender.

SUMMARY:
Befriending services deliver companionship to older adults through regular volunteer visits. ALONE is a charitable organisation providing befriending services to older adults in Ireland. It is the mission statement of ALONE to use befriending to reduce the negative impact loneliness has on health, but evidence for this use of befriending is yet to be sufficiently provided. Providing such evidence would help organisations like ALONE to convince policymakers of the need for, and importance of, their services. The research uses a rigorous scientific approach to evaluate the effect of befriending services on health. Two domains of health thought to be particularly important for ageing adults are evaluated: health-related quality of life (HrQoL), and cognitive function. Maximising HrQoL should be a goal of any healthcare intervention, while cognitive function is associated with dementia risk, a major factor threatening independence in later life. The research is also investigating whether befriending can reduce the negative effect that loneliness is known to have on health of older adults. Service users, befriending volunteers, and professionals involved with the service, will be interviewed by researchers, to see if there are other ways that befriending might improve health. An economic analysis of the service, to evaluate its cost, is also planned. Findings will then be translated all findings into befriending service recommendations for the Department of Health.

To conduct this research, 85 new befriending service users are needed. 10-15 pairs of befriender-befriendees will also be interviewed, and 5-10 health and social care professionals involved with the service. Expected outcomes are to provide ALONE with scientific evidence related to the effects of befriending services on health, and to influence policymakers by clarifying the extent of the economic and health benefits of befriending services.

DETAILED DESCRIPTION:
Background: Loneliness is related to poor health in later life. One way in which loneliness is often addressed is via befriending services, such as those offered by ALONE. The mission statement of ALONE's befriending service is to reduce the impact of loneliness on poor health. ALONE have identified a need for an empirical evaluation of the potential benefits of befriending services. Aims: The proposed research aims to create empirical evidence regarding the impact of befriending services on health and loneliness, assisting ALONE in developing and refining their mission statement. The research question is: "Do befriending services improve health (measured as health-related quality of life and cognitive function), and do they mitigate the impact of loneliness on health?" A secondary aim is to identify, using exploratory methods, potential mechanisms through which befriending impacts health.

Plan of Investigation: A mixed methods design, integrating qualitative and quantitative methods, is planned.

The quantitative component comprises an AB single-case experimental multiple baseline design, analysed using generalised additive modelling, and the qualitative component comprises semi-structured interviews (with befriender-befriendee dyads and healthcare professionals associated with the service) designed and analysed according to the principles of grounded theory. Results will be integrated according to mixed methods guidelines, undergo triangulation, and an economic analysis will evaluate the cost should the service be rolled out nationally. All results will be integrated to form the basis of recommendations for the befriending sector, to be disseminated to policymakers. Results will also be disseminated via peer-reviewed publication and lay report.

Potential Impact: The study has potential to improve the service offered by ALONE by empirically testing its effectiveness and mechanisms of action, influence policy with this information, and contribute to theoretical understanding of the nature of the relationship between befriending, loneliness, and health.

ELIGIBILITY:
Inclusion Criteria:

* being interested in becoming an ALONE befriending service user
* being aged over 60
* having ability to provide informed consent
* having sufficient sensory ability to engage in an interview (if engaging in qualitative component of study)
* self-report of loneliness (responds yes to the question "do you sometimes feel lonely?")

Exclusion Criteria:

* self-report of receipt of a diagnosis by a doctor of any of the following: intellectual disability including autism spectrum disorder or psychotic disorder, dementia, or serious memory impairment
* Living outside the greater Dublin area

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Loneliness | Measured from baseline (point of study registration) and again every two weeks for max. 13 time-points (i.e. 26 weeks in total). At each point of testing, participants are asked to reflect on their loneliness at that point in time.
  University of California at Los Angeles 5-item loneliness scale: This is a five item well validated scale of loneliness suitable for use in older adults. Each item yields scores between 0 and 2. Overall minimum score is 0 and overall maximum score is 10 with higher scores indicating more loneliness.
Change in Health-related quality of life | Measured from baseline (point of study registration) and again every two weeks for max. 13 time-points (i.e. 26 weeks in total). At each point of testing, participants are asked to reflect on their health-related quality of life at that point in time.
  EuroQol 5-Dimension (3-levelL) scale. A well validated scale of health-related quality of life which measures five dimensions of health across three possible levels. Scores can be combined to a summary score which is between 0 (worst health/death) and 1 (best possible health).
Changes in Semantic memory | Measured from baseline (point of study registration) and again every two weeks for max. 13 time-points (i.e. 26 weeks in total).
  Delis Kaplan Executive Functioning System verbal fluency tests standard and alternate: these tests elicit participants' ability to name as many items belonging to a given category (animals, words beginning with F, fruits) as possible in 60 seconds. The minimum value (worst performance) is 0; there is no theoretical maximum value but higher scores indicate better performance.

SECONDARY OUTCOMES:
Changes in Social support | Measured from baseline (point of study registration) and again every two weeks for max. 13 time-points (i.e. 26 weeks in total). At each point of testing, participants are asked to reflect on their social support at that point in time.
  Lubben social network scale (6 item version) - this is a scale which is well validated to be used in older populations and measures social support. Six items ask questions about social support from different sources and scores for each item range from 0-5. The total summed score ranges from a minimum value of 0 (lowest level of social support) to 30 (maximum level of social support).

CONTACTS AND LOCATIONS:
Overall Officials: Joanna McHugh Power, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Trinity College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hannigan C, Hanly P, Kee F, Lawlor B, Holton E, Walsh C, Scharf T, Coen R, Leatham V, Moynihan S, Lane K, McHugh Power J. HALO: Study protocol for a single-case experimental design study evaluating the moderating impact of a befriending intervention on the association between loneliness and health in older adults. HRB Open Res. 2022 Jan 31;3:60. doi: 10.12688/hrbopenres.13104.2. eCollection 2020. PMID 35187395